CLINICAL TRIAL: NCT04325568
Title: Developing Clinical Translational Tools to Communicate Genetic Risk Among Individuals Who Are at Clinical High Risk for Psychosis
Brief Title: Developing Clinical Tools to Communicate Genetic Risk for Individuals Who Are Clinical High Risk for Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R21HG010420 (NIH)
Record Dates: First submitted 2019-10-31; First posted 2020-03-27 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-01

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is a pre-post design (N=54) in which the first 27 participants will take part in the clinician manual intervention and the next 27 participants will be assigned to the AutoTutor. Participants will only complete either the clinical manual intervention or the AutoTutor intervention, but not both. These groups will not be compared to one another. Each participant will be assessed on all outcomes before and after the intervention and will only take part in either the clinician manual or Autotutor. Since each participant is only getting one intervention and the clinician manual and AutoTutor are not being compared to each other the most appropriate study design is single group (and cannot be considered factorial, crossover, parallel, or sequential).
Masking Description: Masking will not be used. Again, the 27 participants will be assigned to the clinician manual and the next 27 participants will be assigned to Autotutor. The investigators are doing this in order to prevent contamination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician Manual (Other): Participants in the Clinician Manual arm will be introduced to a trained clinician and will complete one 60-minute session covering equivalent topics addressed in the PsyGist program. The manual will consist of: (1) a section exploring the youth's causal model for their high-risk state; (2) individualization per their causal model; and (3) tutorials that convey the main concepts of genetic malleability.
  Clinicians will assess individual causal models via discussion with CHR youth about their at- risk state. Individualization of genetic framing will occur using youths' causal models and will fall into 1 of 3 categories (per PsyGist): 'primarily genetic', 'primarily environmental' or 'combined'.
  Interventions: Behavioral: PsyGist and Clinician Manual
- AutoTutor (PsyGist) (Other): AutoTutor is an intelligent system that simulates talking with a human tutor. Our AutoTutor, called PsyGist, has 3 parts: (1) assessment of the youth's causal model for their high-risk state; (2) an individualized 'pre-tutorial' vignette matched to their causal model; (3) a 'tutorial' presenting the 'genetic malleability' framing.
  PsyGist will guide participants through its three components.
  Interventions: Behavioral: PsyGist and Clinician Manual

INTERVENTIONS:
Behavioral: PsyGist and Clinician Manual — This is a pre-post test design aimed at conveying future genetic risk information to those at clinical high risk for psychosis. Participants will be assigned to either complete the Clinician Manual intervention (n= 27 participants) or PsyGist intervention (n=27 participants).

SUMMARY:
While great strides are being made in identifying early signs that place people at a 'high risk state' for different illness conditions, at the same time, advances are being made in the identification of genes associated with 'high-risk states'. This study proposes to develop two innovative clinical tools that could greatly facilitate dissemination of a beneficial genetic malleability framing to high-risk youth in order to encourage increased treatment engagement and uptake of healthy behaviors. The impact of genetic information assumes special importance in the 'high-risk state' because achieving the best possible outcome is more likely if individuals actively choose to engage in beneficial treatment and health-promoting behaviors.

DETAILED DESCRIPTION:
This project seeks to understand how individuals already in a high-risk state will interpret genetic information informing risk of 'conversion' to a full disorder. How individuals interpret this possibility carries important consequences for how they choose to respond, which may range from fatalistic acceptance of the disorder to proactive preventative behavior. With the aim to encourage an active pro-health response, the investigators propose developing two tools for communicating genetic risk and evaluate them regarding their effectiveness in inducing a positive response to the risk of illness. The two tools will consist of: 1) a clinician manual, designed to be used by trained clinicians to communicate risk to CHR youth; 2) a high-impact, computerized tutorial ('AutoTutor') that has been used to convey genetic risk for breast cancer (i.e. BRCA gene). To create these two tools, experts in psychiatric genetics and stigma will work to develop the two tools to convey genetic risk information to youth and young adults identified as in a 'clinical high-risk state' (CHR) for psychosis. The investigators assess primary outcomes of increased intent to engage in treatment and healthy behaviors, and a secondary outcome of reduction in stigma. While specific genes for risk of psychosis are not yet used in diagnosis or treatment, a genetic malleability (GM) framing conforms to the known genetic risk for psychosis, and has a strong likelihood of being used in the not too distant future. Because of the relatively large innovation involved, the investigators seek to establish initial acceptability, safety, and efficacy of each tool. The investigators then use a nonrandomized, within- subject, pre- vs. post design to examine whether providing the genetic malleability framing via each tool (n=27 CHR youth per tool, N=54 total) leads to improved outcomes. For each tool, participants will be conveyed hypothetical information proposing being identified as having a substantially elevated, genetically-malleable risk for developing psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between the ages of 16- 30
* Current or previous COPE participant
* Identified as at clinical high risk for psychosis as defined as having at least one of the following: a)attenuated positive symptoms b)brief intermittent positive symptoms

Exclusion Criteria:

* Meeting CHR via only the Genetic risk and deterioration (GRD) syndrome. If the participant meets the GRD syndrome only, the investigators exclude the rare Genetic risk + deterioration (GRD) syndrome (comprising <1% of CHR cases) because GRD requires having a 1st degree relative with any psychotic disorder, which may be linked with stronger reactions to genetic framings.
* IQ < 80
* Inability to adopt hypothetical situation

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Yang, PhD, Principal Investigator — New York University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician Manual: Participants were introduced to a trained clinician and completed a 60-minute session on genetic counseling material
Period: Overall Study
Arm/Group | Clinician Manual
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants were clinical high risk youth who were in a key period of identity formation.
Arm/Group | Clinician Manual
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 21
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 9
  Gender: Male | 14
  Gender: Other | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 6
  Unknown or Not Reported | 0
Perceived Treatment Efficacy [Mean (Standard Deviation); unit: score on a scale] — Participants rate the likelihood that engaging in treatment and adaptive behaviors reduce the risk for developing psychosis, if they were told they had a genetic risk. Items are measured on a 4-point scale (1=very unlikely, 2=somewhat unlikely, 3=somewhat likely, 4=very likely), with higher scores indicating greater perceived efficacy. Measure is divided into four sub-scales: a) avoiding unhealthy behaviors (4 items range 4-16), b) engaging in healthy behaviors (5 items range 5-20), c) utilizing specialized CHR services (3 items range 3-12), and d) help-seeking behaviors (6 items range 6-24).
  score on a scale
    Avoiding Unhealthy Behaviors | 11.9 (3.2)
    Engaging in Healthy Behaviors | 13.5 (2.8)
    Specialized CHR clinic | 9.6 (1.9)
    Help Seeking | 17.5 (3.3)
Intention to Use Treatment [Mean (Standard Deviation); unit: score on a scale] — Asks participants to rate the likelihood of engaging in treatment and adaptive behaviors, if they were told they had a genetic risk for psychosis. Items are measured on a 4-point scale (1=very unlikely, 2=somewhat unlikely, 3=somewhat likely, 4=very likely), with higher scores indicating greater intention. The measure was divided into four sub-scales: a) avoiding unhealthy behaviors (4 items range 4-16), b) engaging in healthy behaviors (5 items range 5-20), c) utilizing specialized CHR services (2 items range 2-8), and d) help-seeking behaviors (6 items range 6-24).
  score on a scale
    Avoiding unhealthy behaviors | 12.7 (2.9)
    Engaging in healthy behaviors | 13.8 (2.8)
    Specialized CHR clinic | 7.1 (1.3)
    Help Seeking | 17.3 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Perceived Treatment Efficacy
Description: Asks participants to rate the likelihood that engaging in treatment and adaptive behaviors will reduce the risk for developing psychosis, if they were told they had a genetic risk for psychosis. Items are measured on a 4-point scale (1=very unlikely, 2=somewhat unlikely, 3=somewhat likely, 4=very likely), with higher scores indicating greater perceived efficacy. Measure is divided into four sub-scales: a) avoiding unhealthy behaviors (4 items range 4-16), b) engaging in healthy behaviors (5 items range 5-20), c) utilizing specialized CHR services (3 items range 3-12), and d) help-seeking behaviors (6 items range 6-24). Changes in scores from pre- to post-intervention are reported.
Time Frame: Baseline, immediately post-intervention, up to 30 minutes
Population: Participants were clinically high risk youth who were in a key period of identity formation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Manual
Number analyzed (Participants) | 24
score on a scale
  Avoiding Unhealthy Behaviors | 2.6 (2.9)
  Engaging in Healthy Behaviors | 1.6 (2.6)
  Going to a specialized CHR Clinic | 0.5 (1.7)
  Help Seeking Behaviors | 0.5 (2.1)

2. Primary Outcome: Change From Baseline in Intention to Use Treatment
Description: Asks participants to rate the likelihood of engaging in treatment and adaptive behaviors, if they were told they had a genetic risk for psychosis. Items are measured on a 4-point scale (1=very unlikely, 2=somewhat unlikely, 3=somewhat likely, 4=very likely), with higher scores indicating greater intention. The measure was divided into four sub-scales: a) avoiding unhealthy behaviors (4 items range 4-16), b) engaging in healthy behaviors (5 items range 5-20), c) utilizing specialized CHR services (2 items range 2-8), and d) help-seeking behaviors (6 items range 6-24). Changes were measured pre- and post-intervention.
Time Frame: Baseline, Immediately post-intervention, up to 30 minutes
Population: Participants were clinically high risk youth who were in a key period of identity formation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Manual
Number analyzed (Participants) | 24
score on a scale
  Avoiding unhealthy behaviors | 0.9 (1.1)
  Engaging in healthy behaviors | 1.0 (2.4)
  Going to a specialized CHR clinic | -0.3 (1.0)
  Help Seeking behaviors | -0.5 (2.0)

3. Secondary Outcome: Change From Baseline in Self-Stigma About Genetic Risk for Psychosis Development
Description: Assess participants self-stigma if they were told they had a genetic risk for psychosis. 7 items are included: I believe I would be fundamentally different from most people (range 1-4), I would be more likely to do something violent towards other people (range 1-4), I would be more likely to do something violent towards myself (range 1-4), I would be more likely to be unpredictable (range 1-4), I would feel ashamed of myself (range 1-4), I would feel embarrassed about myself (range 1-4), I would think of myself as less competent (range 1-4). each measured on a 4-point scale (1=strongly disagree, 2=somewhat disagree, 3=somewhat agree, 4=strongly agree), with higher scores indicating greater stigma. Change in scores from pre- to post-intervention are reported.
Time Frame: Baseline, Immediately post-intervention, up to 30 minutes
Population: Participants were clinically high risk youth who were in a key period of identity formation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Manual
Number analyzed (Participants) | 24
score on a scale
  I believe I would be fundamentally different from most people | -0.04 (1.0)
  I would be more likely to do something violent towards other people | 0.0 (0.5)
  I would be more likely to do something violent towards myself | 0.2 (0.5)
  I would be more likely to be unpredictable | -0.3 (0.9)
  I would feel ashamed of myself | -0.4 (0.6)
  I would feel embarrassed about myself | -0.3 (0.6)
  I would think of myself as less competent | -0.3 (0.7)

4. Secondary Outcome: Change in Anticipated Discrimination From Others Due to Genetic Risk for Psychosis Development
Description: Assess participants anticipated discrimination if they were told they had a genetic risk for psychosis. 18 items (each with a range of 1-4) are measured on a 4-point scale (1=very unlikely, 2=somewhat unlikely, 3=somewhat likely, 4=very likely), with higher scores indicating greater anticipated stigma. Because this is an exploratory R21 trial, the investigators are also testing and validating new measures for this specific group and purpose however, this is based off a published discrimination scale (Wahl, 1999). Change in scores from pre- to post-intervention for each item are reported.
Time Frame: Baseline, Immediately post-intervention, up to 30 minutes
Population: Participants were clinically high risk youth who were in a key period of identity formation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Manual
Number analyzed (Participants) | 24
score on a scale
  Likelihood of being treated differently by mental health professionals | -0.3 (1.1)
  Likelihood of having trouble keeping or getting a job | -0.4 (0.8)
  Likelihood of being misunderstood by family | 0.0 (0.9)
  Likelihood of being rejected by family | 0.0 (0.7)
  Likelihood of having friends/acquaintances become more distant from you | -0.04 (0.7)
  Likelihood of being targeted by hurtful social media messages | 0.3 (0.7)
  Likelihood of having your friends/acquaintances talk badly about you | 0.1 (0.6)
  Likelihood of having your friends/acquaintances be afraid of you | 0.1 (0.6)
  Likelihood of losing your friends | 0.04 (0.7)
  Likelihood of being looked down on by other people | -0.2 (0.9)
  Likelihood of being overly vigilant that you might become symptomatic | -0.2 (0.7)
  Likelihood of being viewed as someone who is unworthy of trust | 0.0 (0.9)
  Likelihood of being treated as an object of pity | 0.04 (0.8)
  Likelihood of having your insurance status affected | -0.2 (1.1)
  Likelihood of having a school not admit you | 0.04 (0.7)
  Likelihood of having an employer not hire you | 0.2 (1.0)
  Likelihood of having trouble dating | -0.3 (0.9)
  Likelihood of being concerned about having children in the future | -0.3 (0.5)

5. Secondary Outcome: Anticipated Rejection From Others Due to Genetic Risk for Psychosis Development
Description: Assess participants anticipated rejection if they were told they had a genetic risk for psychosis. 3 items (each with a range of 1-4) measured on a 4-point scale (1=very unconcerned, 2=somewhat unconcerned, 3=somewhat concerned, 4=very concerned), with higher scores indicating greater anticipated rejection. Because this is an exploratory R21 trial, the investigators are also testing and validating new measures for this specific group and purpose; however, these items are based off of a published rejection sensitivity scale (Link, Wells, Phelan, Yang, 2015). Change in scores from pre- to post- intervention for each item are reported.
Time Frame: Baseline, Immediately post-intervention, up to 30 minutes
Population: Participants were clinically high risk youth who were in a key period of identity formation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinician Manual
Number analyzed (Participants) | 24
score on a scale
  Scenario 1: Dinner with friends | -0.2 (1.1)
  Scenario 2: Argument with a friend | -0.4 (.8)
  Scenario 3: Dating someone new | -0.1 (1.1)

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Clinician Manual
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04325568/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04325568/ICF_000.pdf